CLINICAL TRIAL: NCT06066047
Title: Low Term Effect of Attentional Touch on Sway Rate Variation of CoP in Asymptomatic Subjects: a Randomized Clinical Trial.
Brief Title: Effect of Attentional Touch in Stabilometric Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accademia Italiana Medicina Osteopatica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 003
Record Dates: First submitted 2023-09-04; First posted 2023-10-04 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Postural Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TOUCH ATTENTIVE TREATMENT (Experimental): 15 minutes of osteopathic treatment with operator's touch attention
  Interventions: Other: TOUCH ATTENTIVE TREATMENT
- AUDITORY ATTENTIVE TREATMENT (Sham Comparator): 15 minutes of osteopathic treatment with operator's auditory attention
  Interventions: Other: AUDITORY ATTENTIVE TREATMENT
- CONTROL (No Intervention): The volunteers lay for 15 minutes in the same environment as the volunteers in the other two groups, without being touched in any way.

INTERVENTIONS:
Other: TOUCH ATTENTIVE TREATMENT — 15-minute treatment using constant touch (0.20 N, approx. 20 grams) developed after training with visual feedback.
  * 5 minutes bilateral touch on external malleolus
  * 5 minutes longitudinal occipital front grip for reciprocal tension membrane movement and Sutherland's fulcrum
  * 5 minutes bilateral touch on acromion, for midline, centring diaphragms
  Throughout the treatment, the practitioner maintained a focused attention on touch by voluntarily and constantly directing attention to the sensation/perception of the hands, perceiving texture, density, temperature, reactivity and motility of the tissue.
  Arms: TOUCH ATTENTIVE TREATMENT
Other: AUDITORY ATTENTIVE TREATMENT — 15-minute treatment using constant touch (0.20 N, approx. 20 grams) developed after training with visual feedback.
  * 5 minutes bilateral touch on external malleolus
  * 5 minutes longitudinal occipital front grip for reciprocal tension membrane movement and Sutherland's fulcrum
  * 5 minutes bilateral touch on acromion, for midline, centring diaphragms
  During the treatment, the operator's attention was focused on acoustic signals delivered through earphones. The beeps were delivered at random intervals between 0.5 and 2.0 seconds. The operator had to count the number of acoustic signals produced during the treatment period.
  Arms: AUDITORY ATTENTIVE TREATMENT

SUMMARY:
Postural balance has been studied in the literature and ideal body mass distribution has been shown to provide stability to the body in an upright position. The use of stabilometry to assess posture is a standard in clinical practice and medical research. In the literature we find osteopathic treatment evaluated with stabilometry in specific pathological conditions. We will experiment on asymptomatic volunteers how attentive touch is effective compared to non-attentive touch and compared to an untreated group by measuring specific parameters that indicate postural balance.

DETAILED DESCRIPTION:
Stabilometry measurements will be taken on asymptomatic volunteers before and after several specific treatments, in particular to measure whether the variance in sway speed is reduced after the treatments. The effect of attentional versus non-attentional touch will be compared in the other two groups, in addition to a control group that receives no treatment.

ELIGIBILITY:
Inclusion Criteria:

• aymptomatics

Exclusion Criteria:

* serious illnesses
* balance disorders
* recent trauma (within 2 years) to the lower limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
the velocity variation of the displacement of the centre of pressure (CoP). | baseline
  The variable is measured with a stabilometric scale (Cyber Sabots) by sampling the signal at 40 Hz.
the velocity variation of the displacement of the centre of pressure (CoP). | 30 minutes
  The variable is measured with a stabilometric scale (Cyber Sabots) by sampling the signal at 40 Hz.

CONTACTS AND LOCATIONS:
Locations (1):
- Studio osteopatico Bettoni, Mantova, Italy